CLINICAL TRIAL: NCT07009106
Title: Improving Postpartum Care Knowledge and Visit Attendance in Expecting Persons With Diabetes Through an Educational Video Pilot Study
Brief Title: Pilot Randomized Control Trial to Assess the Impact of Video Education on Postpartum Care Knowledge and Attendance Among Pregnant Individuals With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Laurie Griffin, Principal Investigator, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1931623
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Postpartum Care
Keywords: Diabetes; Video education
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants received standard prenatal care
- Video Intervention (Experimental): Participants watched a short educational video on postpartum care during a regularly scheduled prenatal visit
  Interventions: Other: Educational video on postpartum care

INTERVENTIONS:
Other: Educational video on postpartum care — Participants watched a short educational video on postpartum care during a regularly scheduled prenatal visit.
  Arms: Video Intervention

SUMMARY:
Each year in the United States, about 700 people die from pregnancy-related causes. More than half of these deaths occur after delivery, during what is often called the "fourth trimester." Many of these deaths-up to 80%-are believed to be preventable. In the first week postpartum, the most common causes of death are heavy bleeding, high blood pressure, and infection. After the first week, heart problems such as cardiomyopathy are the leading causes of death. In addition to the risk of life-threatening complications, health issues like diabetes and high blood pressure during pregnancy can increase a person's risk of developing long-term conditions such as heart disease and type 2 diabetes. Despite the importance of postpartum care, up to 40% of individuals do not attend their postpartum check-up. Attendance is especially low among people who are younger, publicly insured, or from underserved communities. Among individuals with diabetes in pregnancy, postpartum care is critical to monitor blood sugar levels, assess for type 2 diabetes, manage complications, and ensure long-term follow-up with a primary care provider. However, many do not attend this visit or receive recommended screenings. Common reasons include feeling fine, time constraints, and a lack of understanding about the purpose of the visit.

The study was conducted as a pilot randomized controlled trial at a tertiary care center among pregnant individuals with type 1, type 2, or gestational diabetes. Participants were randomly assigned to receive either usual care or to watch a 3-minute animated video during a prenatal visit. After enrolling, all participants completed a baseline survey using a secure platform (REDCap) assessing their knowledge about the postpartum period and care expectations. The video was available in English and Spanish and covered key information about what to expect after delivery, warning signs for complications, and why postpartum care is important. Immediately after viewing the video, participants in the intervention group repeated the knowledge-based questions to assess changes in their understanding. Investigators reviewed the electronic medical records to assess postpartum visit scheduling and attendance. This study is designed to determine whether a brief, accessible educational video can improve postpartum care engagement among individuals with diabetes in pregnancy. If effective, this type of video intervention could be implemented more widely to improve maternal health outcomes, particularly in high-risk populations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 Diabetes, Type 2 Diabetes, or gestational diabetes
* 28 weeks gestational age or later
* 18-50 years of age
* English or Spanish speaking

Exclusion Criteria:

* None

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change in baseline postpartum care knowledge after video education intervention | From pre-video survey during enrollment to immediately after video intervention (1-2 weeks later)
  Among participants randomized to the video intervention group, change in postpartum care knowledge will be assessed using a structured multiple-choice questionnaire administered before and immediately after viewing the educational video on a secure platform (REDCap). Knowledge questions assess understanding of postpartum expectations, complications, and importance of postpartum care. Improvement will be measured by comparing total scores on the pre- and post-video surveys.
Rate of attendance to the postpartum visit | 12 weeks after delivery
  The rate of attendance to a postpartum visit within 12 weeks after delivery will be assessed and compared between groups (video vs. usual care), as documented in the electronic medical record. Attendance will be defined as in-person or telehealth contact with an obstetric provider or primary care provider focused on postpartum care. Differences between groups will be compared using Fisher's exact test.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics & Gynecology Center (OGCC), Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ko JY, Rockhill KM, Tong VT, Morrow B, Farr SL. Trends in Postpartum Depressive Symptoms - 27 States, 2004, 2008, and 2012. MMWR Morb Mortal Wkly Rep. 2017 Feb 17;66(6):153-158. doi: 10.15585/mmwr.mm6606a1. PMID 28207685
- [Background] Kim C, Newton KM, Knopp RH. Gestational diabetes and the incidence of type 2 diabetes: a systematic review. Diabetes Care. 2002 Oct;25(10):1862-8. doi: 10.2337/diacare.25.10.1862. PMID 12351492
- [Background] Thiel de Bocanegra H, Braughton M, Bradsberry M, Howell M, Logan J, Schwarz EB. Racial and ethnic disparities in postpartum care and contraception in California's Medicaid program. Am J Obstet Gynecol. 2017 Jul;217(1):47.e1-47.e7. doi: 10.1016/j.ajog.2017.02.040. Epub 2017 Mar 3. PMID 28263752
- [Background] Attanasio LB, Ranchoff BL, Cooper MI, Geissler KH. Postpartum Visit Attendance in the United States: A Systematic Review. Womens Health Issues. 2022 Jul-Aug;32(4):369-375. doi: 10.1016/j.whi.2022.02.002. Epub 2022 Mar 15. PMID 35304034
- [Background] Galmarini E, Marciano L, Schulz PJ. The effectiveness of visual-based interventions on health literacy in health care: a systematic review and meta-analysis. BMC Health Serv Res. 2024 Jun 11;24(1):718. doi: 10.1186/s12913-024-11138-1. PMID 38862966
- [Background] Bengtson AM, Ramos SZ, Savitz DA, Werner EF. Risk Factors for Progression From Gestational Diabetes to Postpartum Type 2 Diabetes: A Review. Clin Obstet Gynecol. 2021 Mar 1;64(1):234-243. doi: 10.1097/GRF.0000000000000585. PMID 33306495
- [Background] Olerich KLW, Souter VL, Fay EE, Katz R, Hwang JK. Cesarean delivery rates and indications in pregnancies complicated by diabetes. J Matern Fetal Neonatal Med. 2022 Dec;35(26):10375-10383. doi: 10.1080/14767058.2022.2128653. Epub 2022 Oct 6. PMID 36202395
- [Background] Nour NM. An introduction to maternal mortality. Rev Obstet Gynecol. 2008 Spring;1(2):77-81. PMID 18769668
- [Background] Baldwin MK, Hart KD, Rodriguez MI. Predictors for follow-up among postpartum patients enrolled in a clinical trial. Contraception. 2018 Sep;98(3):228-231. doi: 10.1016/j.contraception.2018.04.016. Epub 2018 May 8. PMID 29750924
- [Background] DiBari JN, Yu SM, Chao SM, Lu MC. Use of postpartum care: predictors and barriers. J Pregnancy. 2014;2014:530769. doi: 10.1155/2014/530769. Epub 2014 Feb 20. PMID 24693433
- [Background] Holmes VA, Young IS, Patterson CC, Pearson DW, Walker JD, Maresh MJ, McCance DR; Diabetes and Pre-eclampsia Intervention Trial Study Group. Optimal glycemic control, pre-eclampsia, and gestational hypertension in women with type 1 diabetes in the diabetes and pre-eclampsia intervention trial. Diabetes Care. 2011 Aug;34(8):1683-8. doi: 10.2337/dc11-0244. Epub 2011 Jun 2. PMID 21636798
- See also: CDC — https://www.cdc.gov/hearher/pregnancy-related-deaths/index.html
- See also: ACOG Guidelines — https://www.acog.org/clinical/clinical-guidance/committee-opinion/articles/2018/05/optimizing-postpartum-care
- See also: UptoDate — https://www.uptodate.com/contents/infants-of-mothers-with-diabetes-imd
- See also: March of Dimes — https://www.marchofdimes.org/peristats/data?reg=99&top=5&stop=34&lev=1&slev=4&obj=1